CLINICAL TRIAL: NCT03374397
Title: A Single Center, Randomized, Investigator-initiated Phase III Trial to Evaluate the Efficacy of Preservation of Ovarian Function and Hemostasis, and Its Safety of Surgiguard@ During Laparoscopic Ovarian Cystectomy
Brief Title: PReservation Study of Ovarian Function And Hemostasis, and Its Safety of Surgiguard@ During Laparoscopic Ovarian Cystectomy
Acronym: PRAHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Department of Obstetrics & Gynecology, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1707
Record Dates: First submitted 2017-12-10; First posted 2017-12-15 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Ovarian Cyst Benign
Keywords: Laparoscopic unilateral ovarian cystectomy; SurgiGuard; Hemostasis; Ovarian function preservation; Bipolar electrocauterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SurgiGuard (Active Comparator): Surgiguard Non-woven Drug : SurgiGuard Non-woven 6g during surgery
  Interventions: Drug: Surgiguard
- Bipolar electrocauterization (No Intervention): Bipolar electrocauterization during surgery Drug(-)

INTERVENTIONS:
Drug: Surgiguard — Hemostasis with Surgiguard during laparoscopic unilateral ovarian cystectomy
  Other Names: laparoscopic unilateral ovarian cystectomy
  Arms: SurgiGuard

SUMMARY:
The purpose of this study is to compare hemostasis, ovarian function preservation effect, and safety about intraoperative bleeding with SurgiGuard@ in women who underwent laparoscopic unilateral ovarian cystectomy

DETAILED DESCRIPTION:
In women who underwent laparoscopic unilateral ovarian cystectomy, the effect of SurgiGuard@ was assessed by randomization, using SurgiGuard@ and Bipolar electro cauterization, followed by comparative evaluation of hemostasis, ovarian function preservation, safety using postoperative Hb, anti-mullerian hormone (AMH), pelvis ultrasonography (USG), and physical examination

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years ≤ Ages <45 years
* laparoscopic unilateral ovarian cystectomy scheduled patients with benign unilateral ovarian cyst confirmed by ultrasonography
* women with regular menstruation
* women with regular menstruation cycle from 21 days to 45 days
* Proper state for laparoscopic operation (American society of Anesthesiologists Physical Status classification 1 or 2)
* Patients who signed and approved informed consent

Exclusion Criteria:

* Patients without ovarian cyst
* Patients with malignant female genital disease
* Patients with bilateral ovarian cysts
* Age ≥ 45
* Pregnancy or lactating women
* Serum AMH<0.05 ng/ml
* Patients with endocrine disease such as thyroid abnormality, hyperprolactinemia, cushing disease, etc
* Patients with hormone replacement therapy during 3 months
* Patients who is considered to be difficult to perform the clinical trial when researchers judge

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Hemostasis | post operative 48 hours later,1 week later, and 12 weeks later
  Change of serum hemoglobin from baseline

SECONDARY OUTCOMES:
Ovarian function preservation | post operative 48 hours later,1 week later, and 12 weeks later
  Change of serum AMH from baseline
Volume of ovary | post operative 48 hours later,1 week later, and 12 weeks later
  ovarian volume measured by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park SJ, Seol A, Lee N, Lee S, Kim HS; PRAHA Study Group. A randomized controlled trial of ovarian reserve preservation and hemostasis during ovarian cystectomy. Sci Rep. 2021 Apr 19;11(1):8495. doi: 10.1038/s41598-021-87965-7. PMID 33875738